CLINICAL TRIAL: NCT04988269
Title: COVID-19, Interleukin - 6 and Diurnal Salivary Cortisol
Brief Title: Assessment of Diurnal Salivary Cortisol Production in COVID-19
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Yavropoulou, Senior Endocrinology Consultant, National and Kapodistrian University of Athens
Other Study IDs: Ε.Σ 310
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Adrenal Insufficiency; Adrenal Hyperfunction
Keywords: SARS-CoV-2 infection; Adrenal Cortex; Salivary Cortisol; Salivary DHEA; Aldosterone; ACTH; Interleukin 6; Circadian Rythm
MeSH Terms: conditions — COVID-19; Adrenal Insufficiency; Adrenocortical Hyperfunction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients (Cases): Adult consecutive patients that visited the Emergency Department of LAIKO General Hospital of Athens, Greece from May to July 2021 due to confirmed COVID-19 and related symptomatology.
  Blood sampling on the day of admission (one time point) and saliva sampling at 4 different time points (0.800, 12.00, 18.00,22.00) the next day (all sampling in one day).
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva sampling
- Healthy Controls: Age and gender matched healthy individuals without COVID-19. Blood sampling (at day 1) and saliva sampling at different time points (0.800, 12.00, 18.00,22.00) the next day (all sampling in one day-day 2).
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Saliva sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Assessment of circulating levels of plasma ACTH, plasma aldosterone and serum interleukin -6 levels at day 1
Diagnostic Test: Saliva sampling — Assessment of diurnal variation of cortisol and DHEA levels in the saliva at 4 different time points during the day (0.800, 12.00, 18.00, 22.00) at day 2.

SUMMARY:
In the year of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic several studies have focused on the effect of the COVID-19 on the adrenal cortex, demonstrating conflicting results. Herein, researchers sought to investigate the adrenal response in patients with COVID-19by assessing the diurnal rhythm of salivary cortisol and the adrenal androgen dehydroepiandrosterone (DHEA), as well as the plasma levels of aldosterone and adrenocorticotropic hormone (ACTH) in consecutive patients before the possible therapeutic administration of dexamethasone. To elucidate the potential association between the magnitude of individual immune response and the adrenal cortex response we included serum measurements of interleukin - 6 (IL-6).

DETAILED DESCRIPTION:
All adult consecutive patients that visited the emergency department of the LAIKO General Hospital of Athens from May to July 2021 due to confirmed COVID-19 and related symptomatology were eligible for the study.

Age and gender matched healthy individuals without COVID-19 who had never been treated with GCs and fulfilled the exclusion criteria were also recruited from the Hospital's personnel and included in the analysis as Controls.

Blood samples were obtained immediately upon admission for the measurements of ACTH, IL-6 and aldosterone, which were performed by electrochemiluminescence assays on the cobas e 801 immunoassay analysers (Roche Diagnostics GmbH). Salivary samples for free cortisol and DHEAS were obtained during the next day using the Salivette (Sarstedt, Nümbrecht, Germany) at different time points 0800, 12.00, 18.00, and 22.00. Within 24h after saliva collection the salivettes were centrifuged at 2400 g for 20 min in 4 °C and aliquots were stored at -80 °C and analyzed by an Immunochemiluminescence assay in a Roche COBAS E411 analyzer.

ELIGIBILITY:
Inclusion Criteria:

Adult patients that visited the Emergency Department of LAIKO General Hospital of Athens, Greece from May to July 2021 due to confirmed COVID-19 and related symptomatology

Exclusion Criteria:

(i) pre-existing hypoadrenalism or concurrent systemic glucocorticoid treatment (ii) patients with chronic kidney disease stage 3b and above, (iii) patients with advanced metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital based population. Patients with confirmed COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Diurnal variation of cortisol levels in the saliva (mcg/dL) | One day
  Saliva sampling was performed at 4 different time points during one day (08.00, 12.00, 18.00, 22.00).

SECONDARY OUTCOMES:
Single hormone assessment of plasma ACTH levels (pg/mL) | One day
  Blood sampling was performed on the day of Hospital admission at one time point
Diurnal variation of dehydroepiandrosterone (DHEA) levels (pg/mL) in the saliva | One day
  Saliva sampling was performed at 4 different time points during one day (08.00, 12.00, 18.00, 22.00).
Single hormone assessment of plasma aldosterone levels (pmol/L) | One day
  Blood sampling was performed on the day of Hospital admission at one time point
Single hormone assessment of serum Interleukin-6 levels (IL-6) (pg/mL) | One day
  Blood sampling was performed on the day of Hospital admission at one time point
Single hormone assessment of serum C-reactive protein levels (CRP) (mg/L) | One Day
  Blood sampling was performed on the day of Hospital admission at one time point

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the day of publication and for 1 year.

REFERENCES:
- [Derived] Yavropoulou MP, Filippa MG, Mantzou A, Ntziora F, Mylona M, Tektonidou MG, Vlachogiannis NI, Paraskevis D, Kaltsas GA, Chrousos GP, Sfikakis PP. Alterations in cortisol and interleukin-6 secretion in patients with COVID-19 suggestive of neuroendocrine-immune adaptations. Endocrine. 2022 Feb;75(2):317-327. doi: 10.1007/s12020-021-02968-8. Epub 2022 Jan 18. PMID 35043384